CLINICAL TRIAL: NCT05877742
Title: Around the Turn: A Feasibility Cluster Randomized Controlled Trial of Using Auricular Acupressure to Abstain From Drug Abuse Through Training Nursing Students
Brief Title: AA on Drug Abusers by Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA-drug abusers
Record Dates: First submitted 2023-05-16; First posted 2023-05-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-05

CONDITIONS: Drug Abuse
Keywords: Auricular Acupressure; Nursing Students
MeSH Terms: conditions — Substance-Related Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AA group (Experimental): AA for drug abusers.
  Interventions: Other: AA group
- Control group (Placebo Comparator): Routine seminar for drug abusers.
  Interventions: Other: Control group

INTERVENTIONS:
Other: AA group — Participants will individually receive a 5-minute AA education delivered verbally at his/her respective clinic by a trained nursing student interventionist in addition to the usual scheduled follow-ups and activities at clinics.
  Arms: AA group
Other: Control group — To mimic the time and attention spent, the control group will individually receive a 5-minute seminar delivered by an RA.
  Arms: Control group

SUMMARY:
Drug abuse is a serious public health issue. Despite the serious consequences of drug abuse, there are around 2000 new cases reported by drug abusers each year. There is growing evidence of the use of auricular acupressure (AA), a traditional Chinese medicine (TCM) treatment modality, in reducing withdrawal symptoms among drug abusers. This study aims to investigate the feasibility and effectiveness of training nursing students to deliver brief education on AA on drug abusers.

DETAILED DESCRIPTION:
A 2-arm feasibility cluster RCT will be conducted in the 80 drug abusers from 7 substance abuse clinics in Hong Kong Hospital Authority following the CONSORT statement. The intervention group will receive AA intervention individually from trained nursing students. The control group will individually receive a 5-minute seminar delivered by a research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Have reported to abuse drugs within the past 30 days
* Can communicate in Cantonese and read Chinese

Exclusion Criteria:

* Unstable mental conditions that are not suitable for the intervention
* Receiving acupuncture or acupressure treatment currently or in the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Screening rate | at the 6-month follow-up
  calculated as the number of abusers screened at participated clinics divided by number of abusers at participated clinics during the recruitment period.
Eligibility rate | at the 6-month follow-up
  calculated by dividing the number of abusers who are eligible by the number who are screened.
Consent rate | at the 6-month follow-up
  calculated by dividing the number of abusers who consent to join the study by the number who are eligible.
Randomization rate | at the 6-month follow-up
  calculated by dividing the number of abusers who are randomized into intervention and control groups by those who provide consent.
Attendance rate | at the 6-month follow-up
  calculated by dividing the number of abusers who complete the intervention by those who are randomized.
Retention rate | at the 6-month follow-up
  : calculated by dividing the number of abusers who remain in the study by those who are randomized. Retention rates for the intervention and control groups will be calculated at each follow-up.
Adherence to intervention protocol | at the 6-month follow-up
  calculated by dividing the number of abusers who follow the intervention protocol by those who are randomized.
Complete rate | at the 6-month follow-up
  calculated by dividing the number of abusers who returned questionnaires by the number of questionnaires distributed. This will be calculated by groups at baseline and each follow-up.
Missing data | at the 6-month follow-up
  calculated as the percentage of missing values in the dataset. Unknown or blank values will be considered missing values.
Adverse events | at the 6-month follow-up
  defined as unfavorable and unintended events that are not present at baseline, or appear to have worsened during the study.

SECONDARY OUTCOMES:
Self-reported abstinence | at the 6-month follow-up
  Self-reported drug abstinence at last 30 days.
Abstinence with urine testing | at the 6-month follow-up
  . Those who report no drug abuse within the past 30 days at the 6-month follow-up will be further invited for urine testing.
Self-reported levels of craving | at the 6-month follow-up
  The Chinese version of the 3-item craving scale will be used to measure abusers' self-reported levels of craving.
Anxiety | at the 6-month follow-up
  Generalized anxiety disorder-7 will be used to measure the severity of self-reported anxiety.
Quality of life measures by short-Form Six-Dimension | at the 6-month follow-up
  Short-Form Six-Dimension will be used to assess abusers' quality of life.It contains six dimensions of health. The Chinese version is well validated in Hong Kong.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Principal Investigator — School of Nursing, Hong Kong Polytechnic University
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong